CLINICAL TRIAL: NCT02293538
Title: Evaluation of a Lubricant Eye Drop on Tear Lipid Layer Thickness in Contact Lens Wearers
Brief Title: Formula Identification (FID) 114657 in Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: LCO242-P001
Record Dates: First submitted 2014-11-14; First posted 2014-11-18 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-08

CONDITIONS: Refractive Error
Keywords: Symptoms of Contact Lens Related Discomfort
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 114657 (Experimental): FID 114657 eye drops (10 ml), 1-2 drops instilled in each eye 10 minutes prior to inserting a new pair of habitual contact lenses and after removing them, daily for 2 weeks.
  Interventions: Drug: FID 114657 eye drops (10 ml); Device: Habitual contact lenses
- Saline Control (Active Comparator): Saline control eye drops (15 ml), 1-2 drops instilled in each eye 10 minutes prior to inserting a new pair of habitual contact lenses and after removing them, daily for 2 weeks.
  Interventions: Drug: Saline control eye drops (15 ml); Device: Habitual contact lenses

INTERVENTIONS:
Drug: FID 114657 eye drops (10 ml) — Lubricating eye drop for temporary relief of burning and irritation due to dryness of the eye
  Arms: FID 114657
Drug: Saline control eye drops (15 ml) — Saline eye drops (15 ml)
  Arms: Saline Control
Device: Habitual contact lenses — Commercially marketed biweekly or monthly replacement soft contact lenses as prescribed by eye care practitioner, brand and power

SUMMARY:
The purpose of this study is to evaluate the thickness of the pre-lens tear lipid layer after 2 hours of lens wear with use of FID 114657 compared to saline control.

ELIGIBILITY:
Inclusion Criteria:

* Must sign the informed consent form.
* Stable, tear lipid layer thickness ≤ 75 nm without contact lenses.
* Successfully wearing bi-weekly or monthly replacement soft contact lenses in both eyes for a minimum of 5 days/week during the past 2 months prior to Visit 1.
* Vision correctable to 20/25 Snellen (feet) or better at distance with habitual contact lenses at Visit 1.
* Willing to wear lenses 5 days a week, 8 hours a day for at least 2 days during the study.
* Demonstrate symptoms of contact lens discomfort.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Routinely sleeping in lenses.
* Any active eye inflammation or condition that contraindicates contact lens wear.
* Any systemic diseases that could prevent successful contact lens wear.
* Use of systemic or ocular medications that contraindicate lens wear.
* Fit with only 1 contact lens.
* Unwilling to discontinue the use of cosmetics (such as eyeliner, mascara, or eye shadow) or facial creams on or around the eyelids on Day 1 and Day 14 of the study.
* Women of childbearing potential who are currently pregnant, test positive for pregnancy at Screening visit, breast feeding, or unwilling to use adequate birth control throughout the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Manager, Pharmaceuticals, Global Medical Affairs, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 234 participants were recruited from 6 investigational centers located in the United States.
Pre-assignment Details: Of the 234 enrolled, 84 participants were exited from the study as screen failures and 6 participants were discontinued prior to randomization. This reporting group includes all randomized and treated participants (Intent to Treat) (144).
Groups:
- FID 114657: Formula Identification (FID) 114657 eye drops (10 ml), 1-2 drops instilled in each eye 10 minutes prior to inserting a new pair of habitual contact lenses and after removing them, daily for 2 weeks.
Period: Overall Study
Arm/Group | Saline Control | FID 114657
Started | 73 | 71
Completed | 72 | 69
Not Completed | 1 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants exposed to any test or control article evaluated in this study (Safety Analysis Set). Note: Two participants inadvertently received investigational product without being randomized, so are included in the safety analysis set only.
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline Control | FID 114657 | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (12.25) | 38.3 (12.36) | 36.2 (12.43)
Age, Customized [Number; unit: participants]
  18-64 years | 73 | 71 | 144
  ≥ 65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 65 | 123
  Male | 16 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Mean Pre-lens Tear Lipid Layer Thickness After 2 Hours of Lens Wear on Day 1
Description: The pre-lens tear film is the layer of tears located on top of the contact lens (i.e., between the eye lid and the contact lens). The anterior-most layer of the pre-lens tear film consists of lipids. Lipid layer thickness (LLT) is measured with the LipiView® Interferometer. LLT is measured in interferometric color units (ICUs), where 1 ICU reflects about 1 nanometer (nm) lipid layer thickness. Higher values of LLT indicate a better lubrication of the ocular surface. A thicker tear lipid layer helps reduce evaporation and is indicative of a more stable tear film. The right eye only was used for this measure.
Time Frame: Day 1, after 2 hours of lens wear
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: ICU
Arm/Group | Saline Control | FID 114657
Number analyzed (Participants) | 72 | 71
ICU | 61.2 (21.48) | 61.5 (21.47)

2. Secondary Outcome: Mean Comfortable Lens Wear Time (Time Uncomfortable - Time Insertion) at Baseline and Day 14
Description: At Baseline and on Day 14, comfort was collected through participant questionnaires regarding average and comfortable wear time. Participants filled in what time of day (over the past three days) they usually inserted their lenses, removed them, and at what time they usually became uncomfortable, or if they remained comfortable all day. Comfortable wear time was calculated as Time Uncomfortable minus Time Insertion. The participant rated both eyes together by providing one single rating. This outcome measure was prespecified for only FID 114657.
Time Frame: Baseline (Day 0), Day 14
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FID 114657
Number analyzed (Participants) | 71
hours
  Baseline (n=69) | 7.43 (3.28)
  Day 14 (n=70) | 10.69 (3.53)

3. Secondary Outcome: Percentage of Participants That Experienced At Least 1 Unit Increase From Baseline Score to Day 14 for Overall Comfort With Lenses
Description: Overall comfort was rated by the participant on a 10-point scale, where 1=Poor and 10=Excellent, at Day 0 for their habitual lenses and at Day 14 for the lenses worn for the study during use of the assigned drop regimen. A 1-unit increase indicates improvement. The participant rated both eyes together by providing one single rating.
Time Frame: Baseline (Day 0), Day 14
Population: Intention to treat participants with non-missing observations
Measure: Number; unit: percentage of participants
Arm/Group | Saline Control | FID 114657
Number analyzed (Participants) | 71 | 68
percentage of participants | 84.5 | 79.4

4. Secondary Outcome: Mean Change From Baseline in Comfortable Lens Wear Time (Time Uncomfortable - Time Insertion) to Day 14
Description: At Baseline and on Day 14, comfort was collected through participant questionnaires regarding average and comfortable wear time. Participants filled in what time of day (over the past three days) they usually inserted their lenses, removed them, and at what time they usually became uncomfortable, or if they remained comfortable all day. Comfortable wear time was calculated as Time Uncomfortable minus Time Insertion. A positive change from Baseline indicates improvement. The participant rated both eyes together by providing one single rating.
Time Frame: Baseline (Day 0), Day 14
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Saline Control | FID 114657
Number analyzed (Participants) | 71 | 68
hours | 3.12 (3.72) | 3.28 (3.31)

5. Secondary Outcome: Mean Pre-lens Tear Lipid Layer Thickness After 2 Hours of Lens Wear on Day 14
Description: as for outcome 1
Time Frame: Day 14, after 2 hours of lens wear
Population: Intention to treat participants with non-missing observations
Measure: Mean (Standard Deviation); unit: ICU
Arm/Group | Saline Control | FID 114657
Number analyzed (Participants) | 72 | 69
ICU | 58.5 (21.09) | 59.4 (19.30)

ADVERSE EVENTS:
Time Frame: Reporting of adverse events (AEs) began once informed consent was obtained from the participant, and continued through Day 14. This analysis population includes all participants exposed to any test or control article evaluated in this study.
Description: An Adverse Event (AE) was any untoward medical occurrence in a participant who was administered a study treatment (i.e., initiation of treatment with test article) regardless of whether or not the event has a causal relationship with the treatment. Solicited and spontaneous AE reports were collected for both eyes combined.
Arm/Group | Saline Control | FID 114657
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/72
Other Adverse Events (participants affected / at risk) | 0/74 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.